CLINICAL TRIAL: NCT00237289
Title: Topiramate Versus Placebo as add-on Treatment in Patients With Bipolar Disorder in the Outpatient Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002653
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Bipolar Disorder
Keywords: Manic depression; Mania; Depression; Bipolar disorder; Psychosis
MeSH Terms: conditions — Bipolar Disorder; Mania; Depression; Psychotic Disorders | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to assess the efficacy and safety of adding topiramate as compared to placebo to the medications a patient with bipolar disorder is already taking (lithium or valproate) to see if adding topiramate will better control the patient's manic symptoms.

DETAILED DESCRIPTION:
Many patients with bipolar disorder (manic-depressive illness) require more than one medication to control their symptoms. This is a 12-week, multicenter, randomized, double-blind, placebo-controlled, parallel-groupd study to evalute the efficacy and safety of topiramate versus placebo as add-on therapy to lithium or valproate for the treatment of bipolar 1 disorder as an outpatient setting. These patients must already be taking either lithium or valproate for at least 6 weeks before the first visit and have been on the same dose of the mood stabilizer for at least 2 weeks before the first visit. Paitents will be randomized to receive either placebo or topiramate, an anti-seizure medication not approved for the treatment of bipolar disorder, in addition to their lithium or valporate. The study consists of 56-day titration (topiramate will be titrated up to 400mg per day or the maximum tolerated dose), 28-day continuation period, and 7 days of follow-up to taper off the medication. The study hypothesis is that topiramate will be more effective than placebo in the treatment of mania in type 1 bipolar disorder patients as measured by the Young Mania Rating Scale (YMRS) and will be well tolerated. YMRS is a questionnaire consisting of 11 items designed to assess severity of mania symptoms.

Patients will start taking topiramate 25 mg per day or placebo by mouth. Over the next 8 weeks, doses will be increased to up to 400 mg per day or to the maximum tolerated dose, whichever is lower. After the first 8 weeks, patients will stay at the established dose for the next 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Bipolar Disorder Type I
* Total Young Mania Rating Scale (YMRS) score of 18 or higher
* Currently being treated with a mood stabilizer (lithium or valproate)
* Having a stable therapeutic dose of the mood stabilizer in their bloodstream
* Currently not requiring hospitalization

Exclusion Criteria:

* Patients taking an antidepressant or anti-seizure medication
* Hospitalized paitents
* Women who are pregnant or breast-feeding
* Women who are not using birth control
* Patients with history of drug or alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2001-10; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to final visit in the Young Mania Rating Scale total score. Safety evaluations (incidence of adverse events, physical exams, vital signs, clinical laboratory tests including thyroid function tests) throughout the study.

SECONDARY OUTCOMES:
Changes from baseline to final visit in the Clinical Global Impressions Scale, Global Assessment Scale, Brief Psychiatric Rating Scale, and Montgomery-Asberg Depression Rating Scale. Rate of discontinuation due to efficacy failure.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho McNeil Neurologics, Inc. Clinical Trial, Study Director — Ortho-McNeil Neurologics, Inc.

REFERENCES:
- See also: Topiramate Versus Placebo as Add-On Treatment in Patients with Bipolar Disorder in the Outpatient Setting — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=915&filename=CR002653_CSR.pdf